CLINICAL TRIAL: NCT07025343
Title: Does Intralipid Infusion Can Reverse the Spinal Anesthesia Effect in Day Case Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mahmoud Sharara, MD, Lecturer of Anesthesiology, Intensive Care and Pain Medicine, Faculty of Medicine, Benha University, Egypt., Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 6-1-2025
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Intralipid Infusion; Spinal Anesthesia; Day Case Surgery
MeSH Terms: interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): Patients (>70kg will receive 100 ml, <70 will receive 1.5ml/kg) of 20% intravenous lipid emulsion at the end of surgery as a study group.
  Interventions: Other: Lipid emulsion
- Group C (No Intervention): Patients will not receive intravenous lipid emulsion as a control group.

INTERVENTIONS:
Other: Lipid emulsion — Patients (>70kg will receive 100 ml, <70 will receive 1.5ml/kg) of 20% intravenous lipid emulsion at the end of surgery as a study group.
  Arms: Group S

SUMMARY:
This study aims to evaluate the effect of intralipid infusion on reversing the spinal anesthesia effect in day case surgery.

DETAILED DESCRIPTION:
The increasing demand for day-case surgery has led to a growing interest in developing strategies to provide patients with a more convenient, cost-effective, and less invasive alternative to traditional inpatient procedures.

Spinal anesthesia, in particular, is a widely used technique in day-case surgery due to its ability to provide excellent analgesia with minimal side effects.

Intravenous lipid emulsion therapy is commonly used to treat local anesthetic systemic toxicity (LAST) and has demonstrated some efficacy in treating other drug toxicities, particularly cardiotoxicity from lipophilic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Scheduled for day-case surgery under spinal anesthesia.
* Time of surgery less than 90 min.

Exclusion Criteria:

* Patients with contraindications for outpatient surgery or spinal anesthesia.
* Local anaesthetic (LA) allergy.
* Those receiving anticoagulant therapy.
* Emergency cases.
* Pregnant cases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Onset time of the motor block | Intraoperatively
  The onset time of the motor block using the modified Bromage scale will be assessed. The motor block will be measured when the maximum dermatomal spread is achieved using the modified Bromage scale (0: no motor block, 1: hip blocked, 2: hip and knee blocked, and 3: hip, knee, and ankle blocked).

SECONDARY OUTCOMES:
Duration of motor block | Intraoperatively
  The motor block will be measured when the maximum dermatomal spread is achieved using the modified Bromage scale (0: no motor block, 1: hip blocked, 2: hip and knee blocked, and 3: hip, knee, and ankle blocked).
Time till home readiness | 24 hours postoperatively
  The time to home readiness will be assessed as the time from the end of surgery until the patients reached a post-anesthesia discharge score (PADS) ≥9 and are able to void spontaneously.
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of tramadol administrated).
Total tramadol consumption | 24 hours postoperatively
  Rescue analgesia of 100mg IV tramadol will be given if the numerical rating scale (NRS)> 3 to be repeated after 30 min if pain persists (with maximum dose 400mg) until the NRS < 4.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numerical rating scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable").
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, urinary retention, leg paralysis, or any other complication will be recorded.
Time from the end of surgery till movement | 24 hours postoperatively
  Time from the end of surgery till movement will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Banha University, Banhā, Banha, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.